CLINICAL TRIAL: NCT06240806
Title: Efficacy of Manuka Honey Oral Rinse in Treatment of Xerostomia in Elderly: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Manuka Honey Oral Rinse in Treatment of Xerostomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-061
Record Dates: First submitted 2024-01-14; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Dry Mouth; Salivary Gland Diseases
MeSH Terms: conditions — Xerostomia; Salivary Gland Diseases

STUDY DESIGN:
Intervention Model Description: The experimental group will use a 20ml of (Manuka honey) in 100 ml purified water as mouthwash three times a day (preferably after their meals), kept it for one minute, and then poured it out .
  the control arm followed the same protocol with normal saline rinses in the same opaque bottles 3 times per day.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients in both groups were assigned using a random number table, and then we placed the participants in 2 groups receiving mouthwashes A (Manuka honey) or B (saline oral rinse) based on the randomized list. The researcher, patients, and the statistical analyst were all unaware of which code belonged to which mouthwash and just one non-beneficiary person was aware of the contents of the bottles who revealed them after completing all the statistical analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manuka honey interventional arm (Active Comparator): Manuka honey used as mouth rinse in treatment of xerostomia
  Interventions: Other: Manuka Honey
- Saline mouthwash control group (Placebo Comparator): Saline used as mouth rinse for xerostomia
  Interventions: Other: Saline mouthwash

INTERVENTIONS:
Other: Manuka Honey — Manuka honey will be topically applied to the oral mucosa as oral rinse based on the Biswal et al., 2003 administration protocol.
  Arms: Manuka honey interventional arm
Other: Saline mouthwash — Saline mouthwash will be used 3 times per day for one month
  Arms: Saline mouthwash control group

SUMMARY:
Xerostomia causes many clinical problems, including oral infections, speech difficulties, and impaired chewing and swallowing of food thus may affect the individual's quality of life, therefore this study aimed to evaluate the clinical effectiveness of Manuka honey mouth rinse using the subjective dry mouth score, and patient satisfaction as primary objectives and to assess the effect of Manuka honey on the salivary flow rate, and objective dry mouth score as secondary objectives.

DETAILED DESCRIPTION:
Xerostomia has a variety of possible etiological factors; it is generally classified as having primary and secondary causes. Primary causes comprise conditions that directly affect the salivary glands and induce xerostomia like, Sjogren's syndrome, diabetes mellitus type 1 and 2, thyroid disease, adrenal pathology, renal or hepatic diseases, hepatitis C virus infection, and HIV disease.

Secondary causes of xerostomia include the side-effects of radiation therapy or chemotherapy, rheumatoid arthritis, scleroderma, mixed connective tissues diseases, systemic lupus erythematous, graft versus host disease, anorexia, alcohol and smoking and commonly prescribed drugs (>500 medications reportedly cause dry mouth). The most common medications causing hyposalivation are those with anticholinergic activity, sympathomimetic, and benzodiazepines. The risk of xerostomia increases with the synergistic effects of xerogenic medications, multiple medications, higher doses of medication, and the duration of the medication.

Honey was found to have several benefits as an alternative medicine, it has been used as a natural medicine for more than 2000 years, mainly for wound healing. Though there are many varieties of honey, only some of them e.g. Manuka honey and Malaysian Tualang honey, have been studied in detail for their medicinal properties.

Manuka honey is a monofloral honey, produced from the nectar of flowers of Manuka tree. This variety is produced from the Apis mellifera honey bees, using New Zealand Manuka plants producing specific floral-variety named as Leptospermum scoparium. The composition of Manuka honey consists of carbohydrates, minerals, proteins, fatty acids, phenolic and flavonoid compounds. Although such compounds are found in other types of honey, other unique features also occur in Manuka honey, such as an unusually high level of methylglyoxal (MGO) formed from dihydroxyacetone (DHA) which correlates with antibacterial activity.Manuka honey shows antioxidant and anticancer properties, which are considered due to its constituents-phytochemicals working as active bio-compounds.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders, aged above 65 years.
* All patients must have complaint of xerostomia.
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in subjective dry mouth score | one month
  changes in subjective dry mouth score [Time frame: baseline, 2 weeks, and 4 weeks] after manuka honey mouth rinse use higher number scores mean worse diagnosis while lower values mean better prognosis

SECONDARY OUTCOMES:
Changes in objective dry mouth score | one month
  changes in objective dry mouth score [Time frame: baseline, 2 weeks, and 4 weeks] after manuka honey mouth rinse use higher number scores mean worse diagnosis while lower values mean better prognosis
Increase in Unstimulated Salivary flow rate (ml/min) | one month
  Eating and talking were prohibited during the time of collection. Unstimulated whole saliva was collected for 5 min by spitting method. The collection will be timed, so that flow rate (mL/min) could be measured As the salivary flow rates increased it means improvement
Changes in salivary potential of hydrogen ion (pH) | one month
  following saliva collection, pH was measured immediately using the narrow-range pH strip system (Merck). One drop of the collected saliva was placed on the test strip and its color change reflected the pH of the saliva.
  As salivary pH increased it means improvement

CONTACTS AND LOCATIONS:
Locations (1):
- The British University in Egypt, Cairo, Egypt

REFERENCES:
- [Derived] Ghalwash D, El-Gawish A, Abou-Bakr A. Efficacy of Manuka honey oral rinse in treatment of xerostomia among elderly patients: a randomized controlled trial. BMC Oral Health. 2025 May 23;25(1):777. doi: 10.1186/s12903-025-06125-9. PMID 40410721